CLINICAL TRIAL: NCT00729521
Title: Facilitating Dissemination of Injury Interventions: A Randomized Controlled Trial
Brief Title: Dissemination of Injury Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Peter Layde, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO00007160
Record Dates: First submitted 2008-07-31; First posted 2008-08-07 (Estimated); Results first posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Fall Injury
Keywords: Fall injury hospitalization; Fall injury emergency department visit; Fall injury death

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): a control group receiving no special resources or guidance related to fall injury prevention or the community health improvement process;
- Standard Program (Active Comparator): a "Standard Program" group receiving modest funding to implement an "evidence-based" fall prevention program in their local community;
  Interventions: Other: Standard Program
- Facilitative System (Experimental): a "Facilitative System" group receiving facilitative system support in addition to the resources provided the Standard Program group
  Interventions: Other: facilitative system

INTERVENTIONS:
Other: facilitative system — The facilitative system links communities with academic partners to provide communities with the skills and resources needed to help facilitate the community health improvement process. The system identifies what assets are available within communities, as well as the skills and resources needed to work through the community health improvement process. The facilitative system will then provide technical assistance, best practices guides, and direct consultation in carrying out all phases of the community health improvement process. This information is designed to increase community capacity in community assessment, coalition development, accessing and interpreting local injury prevention data, searching and selecting evidence-based research, and program planning and evaluation.
  Arms: Facilitative System
Other: Standard Program — a "Standard Program" group receiving modest funding to implement an "evidence-based" fall prevention program in their local community;
  Arms: Standard Program

SUMMARY:
An important challenge for the field of injury prevention and control is the translation of research findings into effective community-based prevention programs and practices. The National Center for Injury Prevention and Control believes that dissemination research can overcome this challenge by providing insight into the structures and methods needed to translate injury control research into everyday practice. The proposed dissemination research study will rigorously assess whether the use of a "facilitative system" can successfully bridge the gap between injury prevention and control research and the implementation of evidence-driven, community-based programs, policies, and practices. The facilitative system links communities with academic partners to provide communities with the skills and resources needed to help facilitate the community health improvement process. The system identifies what assets are available within communities, as well as the skills and resources needed to work through the community health improvement process. The facilitative system will then provide technical assistance, best practices guides, and direct consultation in carrying out all phases of the community health improvement process. This information is designed to increase community capacity in community assessment, coalition development, accessing and interpreting local injury prevention data, searching and selecting evidence-based research, and program planning and evaluation. The study will use a randomized community trial design to evaluate fall injury occurrence and process measures of program implementation in three groups of communities:

* a control group receiving no special resources or guidance related to fall injury prevention or the community health improvement process;
* a "Standard Program" group receiving modest funding to implement an "evidence-based" fall prevention program in their local community;
* a "Facilitative System" group receiving facilitative system support in addition to the resources provided the Standard Program group.

We hypothesize that the Facilitative System program will be more effective at:

* reducing fall-related injuries in the elderly;
* building community coalitions that are goal-oriented and sustainable;
* implementing community-based, evidence-driven fall prevention programs that are both tailored to the community needs and yet faithful to empirically-tested fall prevention research studies

ELIGIBILITY:
Inclusion Criteria:

* Communities interested in participating

Exclusion Criteria:

* Existing facilitative system in community

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35037 (Actual)
Dates: Start 2007-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Layde, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 interested communities were randomized to one of the three groups using a block randomization method, taking into account whether the lead agency was a health department or aging agency and whether the community had 0 or 1 or more Stepping On fall prevention program leaders already.
Period: Overall Study
Arm/Group | Control | Standard Program | Facilitative System
Started | 12494 (10 communities in Control with average annual population of 12,494 residents over 65 years old.) | 14842 (Five communities with average annual population of 14,842 residents over 65 years old.) | 7701 (5 communities in Facilitative System with average annual pop. of 7,701 residents over 65 years.)
Completed | 12494 (Average annual population over 65 years old.) | 14842 (Average annual population over 65 years old.) | 7701 (Average annual population over 65 years old.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Average annual population over residents over 65 years of age.
Groups:
- Control: a control group of 10 communities and their residents over 65 years of age receiving no special resources or guidance related to fall injury prevention or the community health improvement process;
- Standard Program: a "Standard Program" group of five communities and their residents over 65 years of age receiving modest funding to implement an "evidence-based" fall prevention program in their local community;
  Standard Program: a "Standard Program" group receiving modest funding to implement an "evidence-based" fall prevention program in their local community;
- Facilitative System: a "Facilitative System" group of five communities and their residents over 65 years of age receiving support in addition to the resources provided the Standard Program group
  facilitative system: The facilitative system links communities with academic partners to provide communities with the skills and resources needed to help facilitate the community health improvement process. The system identifies what assets are available within communities, as well as the skills and resources needed to work through the community health improvement process. The facilitative system will then provide technical assistance, best practices guides, and direct consultation in carrying out all phases of the community health improvement process. This information is designed to increase community capacity in community assessment, coalition development, accessing and interpreting local injury prevention data, searching and selecting evidence-based research, and program planning and evaluation.
- Total: Total of all reporting groups
Arm/Group | Control | Standard Program | Facilitative System | Total
Number analyzed (Participants) | 12494 | 14842 | 7701 | 35037
Age, Categorical [Count of Participants; unit: Participants] — Adults age 65 years.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 0 | 0
    >=65 years | 12494 | 14842 | 7701 | 35037
Sex/Gender, Customized [Number; unit: participants]
  Not collected | NA — Study looked at all older adults over age 65 years and not specifically at male and females | NA — Study looked at all older adults over age 65 years and not specifically at male and females | NA — Study looked at all older adults over age 65 years and not specifically at male and females | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Emergency Department and In-patient Hospitalization for Fall Injury
Description: Rates of fall injury diagnoses per 100 person-years (P-Y) were computed for the communities in each of the study groups for a 2 year baseline period, 2007-2008, and for a 2 year follow-up period corresponding to years 2010-2011. Change in fall injury rates and their 95% confidence intervals (CI) are reported. A mixed-effects Poisson regression model was used to test the presence of an interaction effect on the fall rate between study group and time period (baseline or follow-up). The test is intended to detect a differential time effect by study group. This model, with main effects for study group and time period and an interaction term, will be referred to as the primary model. Model coefficients and incidence rate ratios (IRR) with 95% confidence intervals (CI) are reported.
Time Frame: 2007-2008; 2010-2011
Population: Population of residents aged 65 and older for participating communities in each study arm for 2007-2008 baseline period and 2010-2011 follow-up period.
Measure: Number (95% Confidence Interval); unit: Fall Injury Rate per 100 person years
Arm/Group | Control | Standard Program | Facilitative System
Number analyzed (Participants) | 12494 | 14842 | 7701
Fall Injury Rate per 100 person years
  Fall Injury Rate per 100 P-Y, 2007-2008 | 5.8 [5.7 to 5.9] | 5.9 [5.8 to 6.0] | 6.1 [5.9 to 6.3]
  Fall Injury Rate per 100 P-Y 2010-2011 | 5.8 [5.7 to 5.9] | 5.3 [5.2 to 5.5] | 5.6 [5.4 to 5.8]
Statistical Analysis 1: Comparison: Facilitative System; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Mixed Effects Poisson Regression; Incidence Rate Ratio = 0.92, 95% CI 2-sided [0.88 to 0.95], Standard Deviation 1 — Comparison group is the control arm
Statistical Analysis 2: Comparison: Standard Program; Test type: Superiority or Other; p < .05, Mixed Models Analysis; Mixed Effected Poisson Model Regression; Incident Rate Ratio = 0.91, 95% CI 2-sided [0.88 to 0.94], Standard Deviation 1 — Comparison group is the control arm

ADVERSE EVENTS:
Time Frame: Five years for study period, 2007-2011.
Description: We are not aware of any adverse events associated with this study.
Arm/Group | Control | Standard Program | Facilitative System
Serious Adverse Events (participants affected / at risk) | 0/12494 | 0/14842 | 0/7701
Other Adverse Events (participants affected / at risk) | 0/12494 | 0/14842 | 0/7701

LIMITATIONS AND CAVEATS:
E coding of injuries can be incomplete, but 99.7% of records with a diagnostic code in the range 800-995.89 had an E code. We may have included more than one admission for the same fall, but we excluded admissions from an acute care facility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes